CLINICAL TRIAL: NCT05762224
Title: Comparative Effects of Kinesio Tapping and Pressure Garments on Upper Extremity Lymphedema, Functional Disability and Quality of Life After Mastectomy
Brief Title: Comparative Effects of KT and PG on UE Lymphedema and Functional Disability After Mastectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0547
Record Dates: First submitted 2023-02-20; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Lymphedema of Upper Limb

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effect of kinesio taping on upper limb lymphedema (Experimental): Kinesio taping was applied 2 times a week for 3 weeks to the KT group. KT improves fluid movement by widening the distance between connective tissues like skin and fascia,fascia and muscles and skin and muscles.
  Interventions: Other: Effect of kinesio taping on upper limb lymphedema
- Effect of pressure garments on upper limb lymphedema (Active Comparator): PG group received pressure garments ( 20-60 mmHg)for at least 15 to 18 hours per day for 3 weeks.
  Interventions: Other: Effect of kinesio taping on upper limb lymphedema

INTERVENTIONS:
Other: Effect of kinesio taping on upper limb lymphedema — Group A received Kinesio taping 2 times a week for 3 weeks to reduce lymphedema and Group B received pressure garments(20-60 mm Hg) for at least 15 to 18 hours per day for 3 weeks
  Other Names: USE of Pressure Garments with coventional PT

SUMMARY:
To compare the effects of Kinesio taping and compression garmets on the upper extremity lymphedema,functional disability and quality of life after mastectomy.

DETAILED DESCRIPTION:
The study's primary goal was to find the effects of Kinesio taping and compression garments on the upper extremity lymphedema following mastectomy. This aim was realized through the current study results, the findings of the current study showed that Kinesio taping and compression garments were equally effective on the upper extremity lymphedema following mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* • Age (45 years-75 years)

  * Patients with edema after 1-year mastectomy
  * Unilateral lymphedema
  * Arm circumference change (Arm circumference unilateral than 2 cm or less than 8 cm in comparison with the other side was included)
  * Functional disability or limited movements (shoulder, arm, and hand)

Exclusion Criteria:

* • Active disease leading to swelling

  * Patients on medications, especially diuretics
  * Allergy
  * Infection
  * Pregnancy
  * Heart and kidney diseases
  * Bilateral lymphedema
  * Skin diseases
  * Cellulitis.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2021-12-25 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Girth Measurement (with Tape) | 3 weeks
  The tape was used to assess the limb diameter.
Handgrip strength was evaluated using a dynamometer | 3 weeks
  A dynamometer was used to assess muscle strengthening and hand grip strengthening
The quality of life was assessed by a cancer-specific questionnaire (EORTC QLQ-C30) | 3 weeks
  The EORTC Core Quality of Life Questionnaire (EORTC QLQ-C30) was used to assess the physical, psychological, and social well-being of cancer patients. The EORTC QLQ-C30 was proven to be useful and valid in measuring the quality of life in patients with advanced illness in this investigation
Disabilities of arm, Shoulder and Hand Questionnaire (DASH) | 3 weeks
  The function was assessed using the validated 30-item Quick-Disabilities of Arm, Shoulder, and Hand (Quick DASH) assessment. Respondents are asked to score their capacity to undertake specific activities (such as heavy housework or carrying a shopping bag); the degree of interference with regular social activities, work activities, sleep impairment, pain ratings, and altered sensations

CONTACTS AND LOCATIONS:
Overall Officials: dania sardar, Principal Investigator — Riphah IU; Sobia Kanwal, Study Director — Riphah IU
Locations (1):
- Lahore General Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bao T, Iris Zhi W, Vertosick EA, Li QS, DeRito J, Vickers A, Cassileth BR, Mao JJ, Van Zee KJ. Acupuncture for breast cancer-related lymphedema: a randomized controlled trial. Breast Cancer Res Treat. 2018 Jul;170(1):77-87. doi: 10.1007/s10549-018-4743-9. Epub 2018 Mar 8. PMID 29520533
- [Background] Oliveira MMF, Gurgel MSC, Amorim BJ, Ramos CD, Derchain S, Furlan-Santos N, Dos Santos CC, Sarian LO. Long term effects of manual lymphatic drainage and active exercises on physical morbidities, lymphoscintigraphy parameters and lymphedema formation in patients operated due to breast cancer: A clinical trial. PLoS One. 2018 Jan 5;13(1):e0189176. doi: 10.1371/journal.pone.0189176. eCollection 2018. PMID 29304140
- [Result] Munoz-Alcaraz MN, Perula-de-Torres LA, Serrano-Merino J, Jimenez-Vilchez AJ, Olmo-Carmona MV, Munoz-Garcia MT, Bartolome-Moreno C, Olivan-Blazquez B, Magallon-Botaya R. Efficacy and efficiency of a new therapeutic approach based on activity-oriented proprioceptive antiedema therapy (TAPA) for edema reduction and improved occupational performance in the rehabilitation of breast cancer-related arm lymphedema in women: a controlled, randomized clinical trial. BMC Cancer. 2020 Nov 9;20(1):1074. doi: 10.1186/s12885-020-07558-x. PMID 33167921